CLINICAL TRIAL: NCT04630353
Title: A Phase 0 Trial of HB-201 for Subjects With Transoral Resectable Human Papillomavirus 16 Positive (HPV 16+) Oropharynx Cancer or With Locally Advanced Cervical Cancer Treated With Chemotherapy and Radiation
Brief Title: A Study HB-201 in Patients With Newly Diagnosed HPV16+ Oropharynx or Locally Advanced Cervical Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Hookipa Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-200-002
Record Dates: First submitted 2020-10-23; First posted 2020-11-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-03

CONDITIONS: HPV 16+ Confirmed Oropharynx Cancer and Cervical Cancer
Keywords: HPV; Oropharynx Cancer; Cervical Cancer; Intravenous; Lymphocytic Choriomeningitis Virus; Medical College of Wisconsin Cancer Center; Medical College of Wisconsin; Transoral Surgery; Window of Opportunity; HPV 16+ cervical cancer; HPV 16+ head and neck squamous cell cancer; HPV 16 E7E6; E7E6
MeSH Terms: conditions — Uterine Cervical Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HB-201 Intravenously on Day 1 (Experimental): Patients with resectable stage I-III, HPV 16+ genotype squamous cell cancer of the oropharynx or unknown primary cancer site.
  Interventions: Drug: HB-201 IV
- HB-201 Intravenously 7 to 14 days before chemoradiation (Experimental): Patients with newly diagnosed HPV 16+ genotype advanced cervical cancer, clinical stages IB to IVB with plan for initial treatment of definitive chemoradiation.
  Interventions: Drug: HB-201 IV

INTERVENTIONS:
Drug: HB-201 IV — HB-201 given IV, one (1) time, on day 1.
  Arms: HB-201 Intravenously on Day 1
Drug: HB-201 IV — HB-201 given IV, one (1) time, 7 to 14 days prior to definitive chemoradiation.
  Arms: HB-201 Intravenously 7 to 14 days before chemoradiation

SUMMARY:
This Window of Opportunity clinical trial will examine the immunologic effects of the study agent HB-201 in the head and neck or cervical cancer, when administered by IV route.

DETAILED DESCRIPTION:
The window of opportunity, Study H-200-002, will examine the effects of study agent (HB-201) on subjects during the "window" between diagnosis of their cancer and their definitive cancer surgery or chemoradiation.

The study will be a 2-arm study design. In Arm 1, the study will enroll subjects with resectable stage I-III human papillomavirus 16 positive (HPV 16+) genotype squamous cell cancer of the oropharynx or unknown primary cancer site who are candidates for transoral surgery. Participants will receive a single intravenous dose of the study agent HB-201 prior to transoral surgery administered intravenously.

In Arm 2, the study will enroll cervical cancer subjects who have histologically confirmed newly diagnosed advanced squamous cell carcinoma, adenocarcinoma, and/ or adenosquamous cell carcinoma with HPV 16+ genotype clincal stages IB to IVB with plan for initial treatment of definitive chemoradiation. Participants will receive a single intravenous dose of HB-201 prior to the start of chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Confirmed HPV 16+ (human papilloma virus 16 positive) genotype testing of cancer.
* Disease-free for ≥ 2 years from other curatively treated cancers, with protocol-defined exceptions.
* Evaluated by cardiologist and/or neurologist if protocol-defined cardiac or neurological event within the last 6 months.

HPV 16+ Oropharynx Cancer

* Newly diagnosed, head and neck squamous cell carcinoma or undifferentiated carcinoma of the oropharynx origin or unknown primary cancer site, determined to be resectable.
* AJCC v8.0 Tumor, Node, Metastasis (TNM) stage I-III, cT0- T3, and cervical nodes N1-N3 based on clinical or radiographic criteria with no evidence of distant metastases.
* No prior radiation above the clavicles.
* Must have acceptable renal and hepatic function as defined per protocol.

HPV 16+ Cervical Cancer (Arm 2)

* Newly diagnosed, histologically confirmed advanced cervical cancer (squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma): International Federation of Gynecology and Obstetrics (FIGO) clinical stages IB to IVB with plan for initial treatment of definitive chemoradiation (platinum agent weekly with radiotherapy) for either curative intent or control of local (pelvic) disease.
* No prior radiation to the abdomen or pelvis.
* Must have a safe and accessible tumor lesion amenable for biopsy.
* Must have normal organ and marrow function as defined per protocol.
* Must not have a known allergy to cisplatin, carboplatin, or compounds of similar biologic composition.

Exclusion Criteria:

All subjects:

* Treatment with any systemic anticancer therapy within 3 years (unless agreed otherwise between the Sponsor and the Investigator).
* Treatment with any chronic immunosuppressive medication within 6 months (unless agreed otherwise between the Sponsor and Investigator).
* Uncontrolled diabetes, uncontrolled infection despite antibiotics or uncontrolled hypertension.
* Live vaccine within 28 days (unless agreed otherwise between Sponsor and Investigator).
* Known diagnosis of acquired immunodeficiency syndrome (AIDS).
* Positive Hepatitis B or Hepatitis C tests indicating acute or chronic infection.
* Intercurrent illness likely to interfere with protocol therapy.
* Female subjects who are pregnant or breastfeeding.
* Female subjects of childbearing potential who do not agree to the use of highly effective contraception per protocol.
* Male subjects with sexual partners of childbearing potential who do not agree to the use of protocol-defined contraception

HPV 16+ Oropharynx Cancer (Arm 1)

• Primary tumor or nodal metastasis fixed to the carotid artery, skull base, or cervical spine.

HPV 16+ Cervical Cancer (Arm 2)

* Treatment with chemotherapy for cervical cancer, prior to planned chemoradiation.
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Immune response profiles in subjects with HPV 16+ Head and Neck and cervical cancer. | Approximately 6-8 weeks
  Measurement of antigen-specific CD8+ T cells in blood and tissue (E7E6 antigen specific assay).

SECONDARY OUTCOMES:
Assessment of gene expression and tumor mutational burden (TMB, MSI) in tumor specimens. | Approximately 6-8 weeks
  Pre and post administration of HB-201
Investigate metabolic and proteomics changes in serum and plasma. | Approximately 6-8 weeks
  Pre and post administration of HB-201
Investigate the t-cell receptor repertoire diversity and clonality. | Approximately 6-8 weeks
  Pre and post administration of HB-201.
Clinical evidence of response to HB-201 | Approximately 6-8 weeks
  Change in tumor size per RECIST v1.1
Toxicity profile of HB-201 | Approximately 30 days post HB-201 administration
  Number and type of adverse events per CTCAE v5.0
Other Exploratory Biomarker research may be conducted on any tumor tissue and/or blood samples collected during the study. | Approximately 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Hookipa Biotech GmbH
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No